CLINICAL TRIAL: NCT05910944
Title: European Study of Prodromal iNPH
Acronym: STOP iNPH
Status: Recruiting | Type: Observational
Sponsor: Johan Virhammar (Other)
Collaborators: Swedish Society for Medical Research (Other)
Responsible Party: Sponsor-Investigator, Johan Virhammar, Associate professor, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Other Study IDs: STOP iNPH
Record Dates: First submitted 2023-05-10; First posted 2023-06-20 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Normal Pressure Hydrocephalus; Hydrocephalus
Keywords: natural history; cerebrospinal fluid; biomarkers; long term follow-up
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid Whole blood Plasma Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - prodromal iNPH: Individuals with typical imaging findings consistent with iNPH but none or too mild symptoms to motivate shunt surgery.
  Interventions: Procedure: Shunt surgery
- Group 2 - Healthy controls: Age matched healthy controls
- Group 3 - symptomatic iNPH: Patients with symptomatic iNPH
  Interventions: Procedure: Shunt surgery

INTERVENTIONS:
Procedure: Shunt surgery — Shunt surgery according to each local centers routine
  Groups: Group 1 - prodromal iNPH; Group 3 - symptomatic iNPH

SUMMARY:
To investigate if progression from prodromal into symptomatic NPH can be predicted from advanced neuroimaging, biomarkers in cerebrospinal fluid (CSF) and plasma and investigate the unknown mechanisms causing deterioration by investigating longitudinal changes in the above-mentioned variables. Three different cohorts with both asymptomatic and symptomatic patients as well as healthy controls will be investigated over time, both without intervention and before and after shunt surgery.

DETAILED DESCRIPTION:
Three prospective cohorts will be included during five years from seven European centers.

Group 1 - Prodromal NPH. Patients with imaging features associated with iNPH and no symptoms, or to little symptoms to motivate shunt surgery, will be included prospectively. At baseline, an MRI of the brain will be performed and a lumbar puncture to collect CSF as well as blood samples. The patients will be followed with a standardized scheme that will go on for as long as the patient chose to remain in the study or until the patient develops symptoms and are referred for shunt surgery. The study scheme includes repeated assessments of symptoms, MRI of the brain, CSF samples and blood samples. The following study visits are planned before surgery: baseline, 6 months, 1st year, 2nd year, 4th year, 6th year. After shunt surgery, clinical evaluations and blood samples will be collected at four assessments during five years post-operative.

Group 2 - Healthy controls - For every patient in Group 1, one patient can be included in Group 2. They will be investigated with the same protocol as Group 1 but only follow the protocol for one cycle (Baseline to year 4).

Group 3 - Symptomatic NPH - For each included individual in Group 1 (prodromal NPH), two patients are included in Group 3 (symptomatic NPH). These patients are consecutively included at each centre from routine patients that are planned for shunt surgery. They should be age matched with the individual in Group 1 (+/- 3 years). Their investigations will be identical with the post-operative routine for five years as Group 1.

ELIGIBILITY:
Inclusion criteria - Group 1 - prodromal iNPH

* Brain imaging with both:

  * Evans index > 0.3
  * Callosal angle ≤ 90 º or:
  * Disproportionately enlarged subarachnoid space hydrocephalus (DESH) - defined as: enlarged ventricles, dilated sylvian fissures and tight sulci at the high convexity.
* Absence of symptoms or too mild symptoms to motivate shunt surgery according to local routine, and all of the following:

  * Normal gait pattern, or slight disturbance of the gait pattern that is not considered to be caused by a disease in the central nervous system (CNS).
  * Gait velocity (maximum gait speed), men ≥ 1.4 m/s; women ≥ 1.25 m/s.
  * Rombergs test with eyes open > 60 seconds
  * Mini Mental State Examination (MMSE) ≥ 27 or Montreal Cognitive Assessment (MoCA) ≥ 23
* Informed consent

Exclusion criteria - Group 1 - prodromal iNPH

* Contraindication for MRI
* Other serious disease with expected survival less than three years
* Other type of hydrocephalus:

  * non-communicating hydrocephalus
  * secondary communicating hydrocephalus
  * suspected congenital hydrocephalus (severely enlarged ventricles, narrow sylvian fissures and normal non-compressed sulci at the high convexity or morphological findings consistent with PaVM18)
* Anticoagulants in a dose that hinders lumbar puncture

Inclusion criteria - Group 2 - healthy controls

• Age > 65 years

Exclusion criteria - Group 2 - healthy controls:

* Imaging findings meet inclusion criteria of Group 1
* Previously known relevant neurological disease
* Pathological gait pattern with unknown reason.
* MMSE < 27 or MoCA < 26.
* Anticoagulants in a dose that hinders lumbar puncture

Inclusion criteria Group 3 symptomatic iNPH

* iNPH diagnosis according to international guidelines.19
* Age matched with the individual in Group 1 (+/- 3 years)

Exclusion criteria Group 3 symptomatic iNPH

* Previous stroke (clinical stroke, not only radiologically verified)
* Other serious disease with expected survival less than three years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Group 1 can be included from patients referred to a tertiary hydrocephalus center after investigations/work-up have shown too mild symptoms to motivate shunt surgery.
  Healthy age-matched controls (Group 2) can be included by advertising and by asking relatives to patients in Group 1 and Group 3.
  For each included individual in Group 1 (prodromal iNPH), two patients are included in Group 3 (symptomatic iNPH). These patients are consecutively included at each center from routine patients that are planned for shunt surgery. They should be age matched with the individual in Group 1 (+/- 3 years).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with prodromal iNPH that requires shunt surgery within 6 years from inclusion. | From date of inclusion until decision of shunt surgery, assessed up to 72 months
  Symptoms are assessed with the idiopathic Normal Pressure Hydrocephalus scale (iNPH-scale) with addition of the gait tests: 10 meter walking in maximum speed, timed up and go test (TUG) and 3 m walking backwards. Each center decides when symptoms have progressed enough to motivate shunt surgery according to local traditions and routine. Low values in time and steps of the gait tests indicate good performance and high values of the iNPH-scale (range: 0-100) indicates good performance.
Frequency of patients with prodromal iNPH that progress to symptomatic iNPH | From date of inclusion until 20 points reduction in total iNPH-scale score or 20% reduction in gait speed, assessed up to 72 months
  Symptoms are assessed with the iNPH-scale with addition of the gait tests: 10 meter walking in maximum speed, timed up and go test (TUG) and 3 m walking backwards. A patient is considered symptomatic when total iNPH-scale is reduced by at least 20 points or the mean speed of the gait tests are reduced by 20%. Low values in time and steps of the gait tests indicate good performance and high values of the iNPH-scale (range: 0-100) indicates good performance.
Post operative improvement in iNPH-scale score in patients with mild, moderate and severe preoperative symptoms | Change from preoperative (last visit before surgery) iNPH scale at 3 months, 12 months, 36 months and 60 months follow-up.
  Differences in short (3 and 12 months) and long-term outcome (36 and 60 months) measured as change between preoperative and postoperative iNPH-scale score will be compared between patients with mild, moderate and severe preoperative symptoms. High values of the iNPH-scale (range: 0-100) indicates good performance.

SECONDARY OUTCOMES:
Change in white matter hyperintensities (WMH) | Change from baseline at 24 months, at 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Assess change in volume (mL) of white matter hyperintensities (WMH) measured with volumetric magnetic resonance imaging (MRI) and calculate associations between change in WMH and change in symptoms.
Change in brain morphology | Change from baseline at 24 months, at 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Assess change in brain morphology assessed with the idiopathic Normal Pressure Hydrocephalus (iNPH) Radscale and calculate associations between change in iNPH Radscale and change in symptoms.
Change in ventricular volume | Change from baseline at 24 months, at 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Assess change in ventricular volume (mL) measured with volumetric magnetic resonance imaging (MRI) and calculate associations between change in ventricular volume and change in symptoms.
Change in parenchymal water content | Change from baseline at 24 months, at 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Assess change in parenchymal water content (mL) measured with Synthetic MR and calculate associations between change in parenchymal water and change in symptoms.
Change in cerebral myelin volume | Change from baseline at 24 months, at 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Assess change in cerebral myelin volume (mL) measured with Synthetic MR and calculate associations between change in cerebral myelin volume and change in symptoms.
Changes in plasma biomarkers | Change from baseline at 6 months, 12 months, 24 months, 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Change in plasma levels of neurofilament light chain protein (ng/L), Total-tau (ng/L), amyloid beta-42 (ng/L), glial fibrillary acidic protein (ng/L) will be measured using Quanterix (SIMOA).
Changes in cerebrospinal fluid (CSF) biomarkers | Change from baseline at 6 months, 12 months, 24 months, 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Change in CSF levels of neurofilament light chain protein (ng/L), Total-tau (ng/L), amyloid beta-42 (ng/L), glial fibrillary acidic protein (ng/L) will be measured using Quanterix (SIMOA).
Changes in plasma and cerebrospinal fluid (CSF) proteins | Change from baseline at 6 months, 12 months, 24 months, 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Semi-quantified levels of approximately 200 proteins are measured with proximity extension assay (Neurology panel and Neuro exploratory panel, Olink.com). Measured semi-quantitative in the unit NPX.
Change in quality of life | Change from baseline at 6 months, 12 months, 24 months, 48 months and at time of decision of shunt surgery, assessed up to 72 months
  Quality of life assessed by EQ-5D-5L (EuroQoL 5 Dimensions 5 Levels). A self-assessment questionnaire with five different aspects of quality of life scored on five-level scales.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Virhammar, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (7):
- Kuopio University Hospital, Kuopio, Finland
- Bellaria Hospital, Bologna, Italy
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided